CLINICAL TRIAL: NCT01860261
Title: Pilot Study of the Effects of Exercise on Aging Among Older Persons With HIV
Acronym: SEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UCSF IRB 12-09153
Record Dates: First submitted 2013-04-29; First posted 2013-05-22 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: HIV
Keywords: HIV; AIDS; sedentary; fitness; aging; V02max; d-dimer; IL-6; CRP; ChiWalking; ChiRunning; aerobic exercise; strength training
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic and Strength Training (Experimental): Participants in the Aerobic and Strength Training intervention group will receive a standardized aerobic and strength training exercise program for 12 weeks, including paid gym membership, personal training, and 3 workshops in ChiWalkRun technique.
  Interventions: Behavioral: Aerobic and Strength Training Intervention
- Control (delayed onset of intervention) (No Intervention): After 12 weeks of active observation, this group will receive a modified version of the exercise intervention consisting of a free gym membership for 12 weeks, with limited personal training.

INTERVENTIONS:
Behavioral: Aerobic and Strength Training Intervention — The exercise intervention has three components: (1) aerobic exercise with a metabolic equivalent of task (MET) energy expenditure of at least 900 MET-minutes per week; (2) strength training consisting of 2 sets of 4 upper body exercises (bench press, seated row, shoulder press, and pull down), 3 sets of 3 leg exercises (leg press, extension, and flexion) and 2 sets each of abdominal crunches and back extensions. Weights for each exercise will be gradually increased as participants can complete 12 repetitions for each set on 2 consecutive sessions, with participants performing strength training twice per week total. Three workshops on using ChiWalking or ChiRunning technique for achievement of aerobic activity goals will be provided to participants in the experimental arm.
  Other Names: ChiWalking; ChiRunning
  Arms: Aerobic and Strength Training

SUMMARY:
This pilot study will test the feasibility and acceptability of a 12 week combined aerobic and strength training intervention among persons with HIV who are age 50 or older and do not exercise frequently, and its preliminary effects on aging-related outcomes . The study uses an randomized, controlled trial design and is intended to lead to a larger clinical trial with long-term follow-up. The intervention incorporates small group instruction from a trainer, a small wearable accelerometer to provide accurate data on physical activity, and real-time feedback to participants about exercise levels. The primary outcome measure will be changes in fitness, measured as change in maximal oxygen consumption (VO2 max). The control group will receive a comparable exercise intervention after they complete 12 weeks of observation.

DETAILED DESCRIPTION:
Approximately 40 individuals with HIV infection of at least 6 months duration who currently exercise infrequently will be randomized in a 2:1 ratio to either Intervention Arm (immediate exercise intervention program for 12 weeks duration), or the Control Arm (observation only for 12 weeks duration followed by treatment onset after observation is completed).

Persons assigned to the Intervention Arm will meet initially once per week with a personal trainer, and once per week in small groups with a personal trainer, for a total of two weekly sessions of assisted strength training. In addition, participants will be encouraged to engage in three sessions of aerobic exercise per week of gradually increasing intensity of about 40 minutes duration each, for the 12 week intervention period. Instruction in walking and running form and body awareness that may reduce the risk of injuries (ChiWalking and ChiRunning technique) will be provided to the Intervention Arm by a certified coach during three sessions over the course of the 12 week intervention period as part of the aerobic exercise plan.

Paid gym memberships will be provided for the 12 week treatment period for both groups (memberships for participants assigned to the Control Arm will not begin until the end of the 12 week observation period).

Data will be collected for strength training activity using the passive FitLinxx system at the study gym, and for aerobic steps and pace using accelerometers (Pebble by FitLinxx). Participants in both groups will be asked to wear accelerometers for the duration of the study period.

Participants will be evaluated at baseline, week 6 and week 12 for changes in lab values and questionnaire items. Change in fitness will be assessed using V02 max at baseline and week 12.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Age >=50 years on date of enrollment visit
* Less than 60min/week of vigorous exercise on average in the 90d prior to enrollment
* Able to complete study documents and activities in English (in this pilot we are only prepared to use English language questionnaires and instructional materials)
* Interested in and willing to do an exercise program
* Receiving continuous antiretroviral therapy (ART) for at least six months with an undetectable viral load at most recent clinic visit, or if not on ART then must have been off continuously for six months with no plan to start ART and have CD4 count > 400 cells/µl (to avoid enrolling patients at risk of developing opportunistic infections or other HIV-associated illnesses).

Exclusion Criteria:

* Medical conditions likely to limit the ability to participate in the planned exercise, including renal failure (creatinine > 2 mg/dl, congestive heart failure, significant lung disease, or severe osteoarthritis, Any health condition(s) that the study physician determines would preclude safe participation in the intervention or may require special modification of the exercise protocol (e.g. angina or myocardial infarction in the past 6 months)
* Substantial deconditioning or current impairment of physical function; this will be tested for by assessing whether patients can climb up and back down one flight of stairs (approximately 3 meters of elevation gain) without stopping 8.
* Unable or unwilling to actively participate in the intervention for the duration of the pilot study
* Unable to provide informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
VO2 max | 12 weeks (baseline to exit)
  Fitness will be assessed by maximal oxygen consumption (V02max) during a stationary bike test, to be completed at baseline and repeated 12 weeks later at the exit visit.

SECONDARY OUTCOMES:
METs | 12 weeks (baseline to exit)
  The measure will assess change in physical activity as summarized by METs (metabolic equivalent tasks), as measured by an accelerometer. Accelerometer data will be available for both the intervention and control groups.
C-reactive protein | Six weeks (baseline to week 6) and 12 weeks (baseline to exit)
  The investigators will assess change in high-sensitivity C-Reactive Protein using blood samples drawn and processed at baseline, week 6 (interim) and week 12 (exit).
NIH PROMIS 29 | 6 weeks (baseline to week 6) and 12 weeks (baseline to exit)
  NIH PROMIS-29 Adult Profile measures will be collected by computerized self-assessment or paper questionnaire. These will include current depression and anxiety, physical functioning and mobility, fatigue, sleep, pain, and ability to participate in social roles and activities (this is a standardized instrument in NIH PROMIS called "The PROMIS-29 Adult Profile"). These data will be collected at baseline, week 6 (interim) and week 12 (exit) for both intervention and control groups.
Feasibility of recruitment | 11 weeks (01Jan2013 to 14Mar2013)
  The investigators will determine how many persons must be screened and enrolled in order to complete cohort enrollment targets.
Acceptability of study materials | Six months (01Jan2013 - 30June2013)
  The investigators will assess the appropriateness and quality of study procedures from the point of view of the study participants. To do this, they will collect questionnaire data. Key procedures (such as V02max, use of the accelerometer) will be rated as "highly acceptable", "acceptable/could be improved" or "needs improvement".
Average distance walked/run per week | From baseline to week 12
  The average change in distance traveled by walking or running per week, as measured by an accelerometer, from the beginning of the study until week 12 will be compared between treatment groups.
Injuries | From study baseline to week 12
  Exercise related injuries, from self-report on questionnaires, will be compared between groups.
Self-reported physical activity | Change from week 0 to week 12
  Change in self-reported physical activity levels, as average minutes of physical activity of different intensity levels, will be compared between groups using the International Physical Activity Questionnaire (IPAQ).

OTHER OUTCOMES:
CD4+ T-cell count | change from week 0 to week 12
  Change in CD4+ T cell counts during the intervention will be compared between groups.
d-dimer | change from week 0 to week 12
  If funding permits, change in d-dimer will be compared between groups form week 0 to week 12.
CD4 cluster of differentiation 4 Other Pre-Specified Outcome Measure IL ileum immature lung independent laboratory inguinal ligament interleukin (IL)-6 | week 0 to week 12
  If funding permits, change in IL-6 will be compared between groups, from week 0 to week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M Hecht, M.D., Principal Investigator — UCSF Osher Center for Integrated Medicine, UCSF Positive Health Program
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States